CLINICAL TRIAL: NCT06373432
Title: Intrapartum Glucose Monitoring of GDM: A Randomized Controlled Trial
Brief Title: Frequency of Glucose Monitoring in Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Thomas Owens, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY-22-01607
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Neonatal Hypoglycemia

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infrequent testing (Experimental): Finger sticks every 4 hours in latent labor (less than 5cm cervical dilation) and every 2 hours in active labor (6cm and greater)
  Interventions: Other: Fingerstick
- Frequent testing (Placebo Comparator): Finger sticks every 2 hours in latent labor (less than 5cm cervical dilation) and every 1 hours in active labor (6cm and greater)
  Interventions: Other: Fingerstick

INTERVENTIONS:
Other: Fingerstick — Fingerstick to check glucose value during labor.

SUMMARY:
The aim of this study is to assess rates of neonatal hypoglycemia with differing intrapartum glucose protocols. Currently at this time there is no guidance from professional medical organizations about when and how frequent to assess maternal glucose levels intrapartum. Several institutions have no protocols in place. The study will be a randomized controlled trial placing patients with Gestational Diabetes Mellitus (GDM) in "frequent" vs "infrequent" glucose monitoring intrapartum and assessing neonatal glucose levels at birth.

ELIGIBILITY:
Inclusion Criteria:

* All female patients of reproductive age who have the diagnosis GDM
* Patient with singleton gestation presenting in labor or for induction

Exclusion Criteria:

* Patients below the age of 18
* Multiple gestation pregnancy
* Patients undergoing scheduled c-section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Neonatal Hypoglycemia | end of study at 6 months
  Glucose values of neonate measured in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Owens, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No